CLINICAL TRIAL: NCT02005224
Title: Effect of Low-carbohydrate/High-fat Diet on Glucose Tolerance and Lipid Profile in Lean, Healthy Women
Acronym: LCHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantis Medical University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMUC-NIH-LCHF-P1-2012
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Insulin Sensitivity; Weight
Keywords: Insulin sensitivity; Lipid profile; Body composition; Weight
MeSH Terms: conditions — Insulin Resistance; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LCHF diet and a bout of exercise (Other): LCHF diet for 3 weeks, where E% 70 fat, E% 20-25 proteins and 20g or less carbohydrates. Oral glucose tolerance test on the morning of day 21 followed by a bout of exercise in the afternoon (indoor bicycle, 60min at 75% HFpeak). The following morning (day 22) a new oral glucose tolerance test. Oral glucose tolerance test results from pre-tests used to determine the effect of LCHF and a bout of exercise on insulin sensitivity.
  Interventions: Other: LCHF diet and a bout of exercise

INTERVENTIONS:
Other: LCHF diet and a bout of exercise — Low-carbohydrate/high-fat diet; effect on insulin sensitivity, lipid profile, weight and body composition. Participants ingested LCHF diet for three weeks before undergoing an oral glucose tolerance test. The same afternoon the participated in an one hour indoor bicycle training at 75% at HFpeak. The following morning they underwent a new oral glucose tolerance test. Body composition and weight were measured before and after the intervention. Oral glucose tolerance test was also performed before the intervention for baseline. Blood samples were collected before and after the intervention for lipid profile analyses.

SUMMARY:
Intervention studying the effect of a low-carbohydrate/high-fat (LCHF) diet as well as on bout of exercise in combination with either a normal diet or a LCHF diet, in relation to glucose metabolism, insulin sensitivity, lipid profile and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Normal weight
* BMI between 18.5 and 25
* Moderately trained

Exclusion Criteria:

* Smokers/tobacco users
* pregnancy
* familial cardio-vascular-disease
* diabetes or reduced glucose tolerance
* under- or overweight (BMI under 18.5 or over 25)
* top athletes

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve glucose (0, 15, 30, 45, 60, 90 and 120 min) | -1 week, 3 weeks
  performed by oral glucose tolerance test, 75 g glucose, 300 ml water

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen Jensen, PhD, Study Director — Norwegian School of Sport Sciences - Department of Physical Performance
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway